CLINICAL TRIAL: NCT05529680
Title: Impact of Scapular Mobilization And Strengthening Exercises on Shoulder Function Post Mastectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Shaimaa Mohamed Ahmed Elsayeh, Lecturer of physical therapy, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P.T.REC/012/003464
Record Dates: First submitted 2022-09-02; First posted 2022-09-07 (Actual); Last update posted 2022-09-07 (Actual); Status verified 2022-09

CONDITIONS: Oncologic Complications; Exercise Therapy; Shoulder Pain; Shoulder Syndrome
Keywords: Scapular mobilization; Scapular strengthening exercises; Mastectomy; Shoulder function
MeSH Terms: conditions — Shoulder Pain

STUDY DESIGN:
Intervention Model Description: Forty patients suffering from post-mastectomy shoulder dysfunction were randomly assigned into two equal groups each one has 20 patients.
  Group A (study group): Who received scapular mobilization and strengthening exercises in addition to their conventional physical therapy program.
  Group B (control group): Who received a conventional physical therapy program in form of joint mobilization, posterior capsule stretching, and range of motion exercise.
Who Masked: Participant
Masking Description: the patients were randomly assigned into two equal groups (20 patients for each group) by using the closed envelope method.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Scapular mobilization and strengthening exercise (Experimental): Group A (study group):
  This group included 20 patients with shoulder dysfunction post-mastectomy who received scapular mobilization and strengthening exercise in addition to their conventional physical therapy program in form of joint mobilization, posterior capsule stretching and range of motion exercise (ROM).
  Interventions: Other: Scapular mobilization and Scapular strengthening exercises; Other: Conventional physical therapy program
- Conventional physical therapy program (Active Comparator): This group included 20 patients with shoulder dysfunction who received conventional physical therapy programs in form of joint mobilization, posterior capsule stretching, and range of motion exercise (ROM).
  Interventions: Other: Conventional physical therapy program

INTERVENTIONS:
Other: Scapular mobilization and Scapular strengthening exercises — The intervention was applied for four weeks, 3 sessions/week. and the Shoulder Pain and Disability Index (SPADI): for measurement of shoulder disability and the Inclinometer: for measurement of shoulder flexion, abduction, external rotation, and scapular upward rotation were used for shoulder assessment before and after the intervention for both groups.
  Arms: Scapular mobilization and strengthening exercise
Other: Conventional physical therapy program — The intervention was applied for four weeks, 3 sessions/week. and the Shoulder Pain and Disability Index (SPADI): for measurement of shoulder disability and the Inclinometer: for measurement of shoulder flexion, abduction, external rotation, and scapular upward rotation were used for shoulder assessment before and after the intervention for both groups.

SUMMARY:
The most common complications following mastectomy are pain, lymphedema of the upper limb ipsilateral to surgery, decreased range of motion (ROM), limited to 90° of flexion, abduction, and external rotation to 40° of the shoulder, and postural changes. It was reported that 60% of breast cancer patients show a reduction in shoulder flexion and abduction at 1-month post-surgery and 10% of survivors show a persistent ROM reduction at 12 months. So, The purpose of the study was to evaluate the therapeutic impact of scapular mobilization and strengthening exercises on shoulder function post-mastectomy.

DETAILED DESCRIPTION:
In this randomized controlled trial study (RCT), forty female patients "The patient's ages ranged from 40 to 55 years" suffering from post-mastectomy shoulder dysfunction ((20° ≥ ROM limitation compared to the sound shoulder & 3 months to 6 months post mastectomy) were randomly assigned into two equal groups, each one had 20 patients.

Group A (study group): This group included 20 patients with shoulder dysfunction post-mastectomy who received scapular mobilization and strengthening exercise in addition to their conventional physical therapy program for four weeks, three sessions/week.

Group B (control group): This group included 20 patients with shoulder dysfunction who received conventional physical therapy programs in form of joint mobilization, posterior capsule stretching, and range of motion exercise (ROM) for four weeks, 3 sessions/week.

Equipment and tools:

* Measurement tools were (The shoulder Pain and Disability Index (SPADI): for measurement of shoulder disability and inclinometer: for measurement of shoulder flexion, abduction, external rotation, and scapular upward rotation), the measurements were recorded before and after the study.
* Therapeutic equipment and tools were (Thera Bands of different colors and resistance and dumbbells of different weights).

The potential participants were excluded if they met any of the following criteria: Diseases such as rheumatoid arthritis, history of trauma or accidental injuries, neurological involvement (stroke, Parkinsonism), history of surgery on the involved shoulder, and diabetic patient.

ELIGIBILITY:
Inclusion Criteria:

* Female patients with ages ranging from 40-55 years.
* All patients had shoulder dysfunction post-mastectomy (20° ≥ ROM limitation compared to the sound shoulder).
* Patients were 3 months to 6 months post-mastectomy.
* All enrolled patients signed the informed consent.

Exclusion Criteria:

* Disease such as rheumatoid arthritis.
* History of trauma or accidental injuries.
* Neurological involvement (stroke, Parkinsonism).
* History of surgery on the involved shoulder.
* Diabetic patient.

Ages: 40 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — female patients
Enrollment: 40 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2022-06-28 (Actual); Study Completion 2022-07-20 (Actual)

PRIMARY OUTCOMES:
Changes in Inclinometer reading before and after the treatment. | Baseline and four weeks after the intervention
  for measurement of shoulder flexion, abduction, external rotation, and scapular upward rotation
Changes in Shoulder Pain and Disability Index (SPADI) before and after the treatment. | Baseline and four weeks after the intervention
  for measurement of shoulder disability

CONTACTS AND LOCATIONS:
Overall Officials: Shaimaa Elsayeh, PhD, Study Director — Cairo University
Locations (1):
- Shaimaa Mohamed Ahmed Elsayeh, Cairo, New Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No